CLINICAL TRIAL: NCT07076511
Title: A Novel, Intuitive Airway Trolley to Facilitate Fast Decision Making in the Emergency Scenario "Unexpected Difficult Airway": Evaluation and Comparison to the Existing Airway Trolley in the Scope of a Simulation Training
Brief Title: A Novel Intuitive Airway Trolley for Quick Decision-making in Simulated Unexpected Difficult Airway Situations: Evaluation and Comparison to the Existing Airway Trolley
Acronym: Airway-to-Go
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Katharina Epp, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Airway-to-Go
Record Dates: First submitted 2023-07-16; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Airway Morbidity; Team Efficacy; Intubation; Difficult or Failed; Human Factors
Keywords: Difficult Airway Trolley; Human factors; Team performance; visual aids

STUDY DESIGN:
Intervention Model Description: randomized, controlled, single-blinded simulation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel Airway Trolley (Active Comparator): Participants are asked to solve a scenario "unexpected difficult airway" using the novel Airway Trolley with color-coding and visual aids
  Interventions: Other: Scenario "unexpected difficult airway"
- Existing Airway Trolley (Placebo Comparator): Participants are asked to solve a scenario "unexpected difficult airway" using the existing Airway Trolley without color-coding and visual aids
  Interventions: Other: Scenario "unexpected difficult airway"

INTERVENTIONS:
Other: Scenario "unexpected difficult airway" — Participants are asked to solve a scenario "unexpected difficult airway" using a manikin in accordance with current guidelines. The scenario aims for participants to try 3 different techniques in securing the airway before performing emergency front of neck access.

SUMMARY:
The goal of this study is to analyze the impact of color-coded labeling and cognitive visual aids of a novel airway trolley on the performance of participants in a simulated unexpected difficult airway scenario. All participants will complete the same scenario, randomized to either the novel or the existing airway trolley. The main questions aimed to be answered are:

1. how long does it take to solve the scenario (=establish sufficient oxygenation via emergency front of neck access) with the novel vs the existing airway trolley?
2. how many deviations from the algorithm "unexpected difficult airway" are documented for each trolley (novel vs existing)?
3. are there differences in the provider experience between both trolleys

ELIGIBILITY:
Inclusion Criteria:

* anaesthesiological 2nd and 3rd year residents at University Medical Centre Mainz
* anaesthesiological attendings at University Medical Centre Mainz
* informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Time to emergency front of neck access (eFONA) decision (in s) | time (in seconds) until scenario is solved and decision to perform eFONA is verbalized (maximum time to solve scenario 10 minutes)
  time to verbalized decision to perform eFONA defined as time to solving the scenario (in s)

SECONDARY OUTCOMES:
Time to decision to prepare eFONA (in sec) | time (in seconds) when decision to prepare eFONA is verbalized (maximum time to solve scenario 10 minutes)
  Time until the decision to prepare (but not directly execute) eFONA (in sec)
Time to establish successful oxygenation (in seconds) | Maximum time to solve scenario: 10 minutes
  Time to establish successful oxygenation (defined as successfully conducting eFONA and performing ventilation) in seconds
number of departures from difficult airway algorithm | Through the course of the scenario (maximum time for completion 10 minutes)
  The number of times during the scenario that the treatment is not concordant with the difficult airway algorithm
Gender differences in the time until eFONA | Maximum time to solve the scenario: 10 minutes
  Gender differences in the time until eFONA is performed
Gender differences in number of departures from difficult airway algorithm | Maximum time to solve the scenario: 10 minutes
  Gender differences in number of departures from difficult airway algorithm
subjective work load evaluation | To be filled out after completing the scenario (time given: 3 minutes)
  evaluating the work load using NASA task load scale (NASA-TLX) questionnaire (nominal scale from very low to very high)
number of unnecessary drawer opening | Through the course of the scenario (maximum time for completion 10 minutes)
  The number of times during the scenario that drawers are opened without retrieving any equipment
subjective operator experience | To be filled out after completing the scenario (time given: 3 minutes)
  Experience of the operator using an ordinal scale (1-7)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, University Medical Centre of Johannes Gutenberg University, Mainz, Rhineland-Palatine, Germany

IPD SHARING:
Plan to Share IPD: Undecided